CLINICAL TRIAL: NCT04717232
Title: Effectiveness of Interprofessional Mentoring Competence Education for Dental Health Care Professionals: A Quasi-experimental Study Protocol
Brief Title: Effectiveness of Interprofessional Mentoring Competence Education for Dental Health Care Professionals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Anna-Leena Keinanen, Principal Investigator, University of Oulu
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: MentoringComperence
Record Dates: First submitted 2020-12-16; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Competence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The blended learning approach to mentoring education for dental health care professionals (Experimental): The blended learning approach to mentoring education for dental health care professionals will last five weeks, including four face-to-face seminars, interprofessional group work and self-reflection assignments lasting for two days. The educational content will include mentoring as a process, mentoring as a relationship, challenges of mentoring, and personal mentoring.
  Interventions: Other: Blended learning approach to mentoring education for dental health care professionals
- The interprofessional online mentoring education (Experimental): The intervention group will attend mentoring competence education. The Interprofessional online mentoring educations includes videos of specialist lectures, e-learning materials, along with assignments concerning reflection skills and participant-based evaluation. The education content included the processes and interactions of mentoring, goal-oriented mentoring, along with student-based feedback and student-centered evaluation. The mentoring education can be completed in an online learning environment and participants can complete the education at their own pace within six weeks.
  Interventions: Other: The interprofessional online mentoring education
- The Control group (Active Comparator): The control group are dentists´ and dental hygienists´ who are working at health care centers on the Finnish Dental Association site, participate in student mentoring and have not received any education before.
  Interventions: Other: Blended learning approach to mentoring education for dental health care professionals; Other: The interprofessional online mentoring education

INTERVENTIONS:
Other: Blended learning approach to mentoring education for dental health care professionals — The participants in the intervention group are dentists´ and dental hygienists´. The mentoring education for dental health care professionals (3 ECTS credits) will be organized by the program leader in Dentistry at the place-blinded. The aim of the mentoring education is to build understanding of how to support a student's professional development (both basic education and specialization) and transfer skills that are relevant to working as an independent expert in oral health care.
  Arms: The Control group; The blended learning approach to mentoring education for dental health care professionals
Other: The interprofessional online mentoring education — The participants in the intervention group are dentists´ and dental hygienists´. The interprofessional online mentoring education (3 ECTS credits) will be organized in collaboration with the Finnish Dental Association in an online environment. The aim of the intervention is to in-crease mentors' competence in guidance processes and interactions, supporting students´ goal-oriented learning and professional evaluation, and providing constructive feedback.
  Arms: The Control group; The interprofessional online mentoring education

SUMMARY:
Clinical practice is an integral part of dental and dental hygiene students' education. The curriculum for a degree is guided by best academic practices for European undergraduate dental education, published by the Association for Dental Education in Europé (ADEE), and the dental hygienist education is based on a European qualifications framework. Interprofessional education has been recognized as a means to improve oral health professional training due to the linked form of education with improved health outcomes.

The interprofessional mentoring education is needed for the clinical practice, which has to be implemented in interprofessional teams. Clinical practice mentors need to have completed an interprofessional mentoring education. Different types of educational approaches have been previously affecting mentors' competence development in mentoring. Dental and dental hygiene students can experience team-based, interprofessional education by participating in clinical practice sessions offered in a communal learning environment. Traditional lectures can be transformed into modern, enhanced learning experiences that correspond to the new generation of students. Online learning methods are increasingly being incorporated into dental health care education. Online learning is designed to be able to support learners with technology supporting and facilitating student learning. Those methods can be used in dental health care continuous education.

This study is designed to evaluate educational intervention's effectiveness of inter-professional mentoring education on mentors' competence development of dentists and dental hygienists mentors.

DETAILED DESCRIPTION:
METHODOLOGY

Study setting:

The interprofessional intervention applying blended learning will be conducted at the higher education institution's interactive learning facilities, while the online interprofessional intervention will be conducted in an online learning environment in collaboration with the teaching-learning company of the Finnish Dental Association.

Study design:

This is a nonrandomized pre-post quasi-experimental study. The participants in this study will participate in interprofessional mentoring education. Participants will self-assess their level of Competence in mentoring, which includes seven dimensions; mentor characteristics, mentor motivation, mentoring practices in the workplace, reflection during mentoring, goal-oriented mentoring, student-centered evaluation and constructive feedback. There will be three assessment time points: at baseline (before education, T0), immediately after the education (T1), and 3 months after the education (T2). The control group will not receive any educational intervention. The interventions and control group will be used the same self-assessment instrument and assessment time points.

Study size:

The intervention and control groups will include 60 participants per group. The 60 participants in the intervention group will be further divided into two groups: one group (30 participants) completing the blended learning module and the other group (30 participants) completing an online learning module.

Study duration:

The intervention will be conducted for a duration of 6 months. More precisely, the blended learning module will be offered twice, in spring 2019 and spring 2020. The online learning module will be conducted during spring 2020 and autumn 2021.

Sampling of participants

Recruitment:

An announcement about both interventions will be published in Finnish journals of dental health care and the official journal of the Finnish Dental Association. The mentors can then choose which form of education was more convenient in terms of time and location. The blended learning approach will be offered once per year in the springtime, while the online mentoring education is available throughout the year.

Intervention:

Blended learning approach to mentoring education for dental health care professionals for participants (dentists and dental hygienists) in the intervention group comprises completion of specialist lectures, discussions, interprofessional group work and self-reflection. The mentoring education will last five weeks, include four face-to-face seminars (2+2 days) and self-reflection assignments lasting an estimated two days.

The online mentoring education for participants (dentists and dental hygienists) in the intervention group comprises of completion of represents a collaboration between members of the dental association, specialist lectures and the coordinator of the dental association. The online mentoring education environment, Priima, includes videos of specialist lectures, e-learning materials, along with assignments concerning reflection skills and participant-based evaluation. In addition, the learners will be informed that they could get in touch with the coordinator of the association if necessary.

Control:

The participants in the control group are dentists and dental hygienists who are listed as working at health care centers on the Finnish Dental Association site (tkharjoittelu.hammaslaakariliitto.fi) and participate in student mentoring. Data concerning the control group, which did not receive any educational intervention. The control group represents dentists or dental hygienists from randomly selected organizations, while all of the participants will be selected from subdivisions of the 2007 NUTS (Nomenclature of Territorial Units for Statistics). Control group randomization will be performed via Research Randomizer (https://www.randomizer.org/#randomize) and ensured that participants in the intervention groups are similar with respect to both known and unknown prognostic factors.

Sample size:

The target of participant selection is to obtain a sufficiently large sample size that represents a highly heterogeneous study group so that concrete conclusions about the effectiveness of the educational interventions can be drawn. A power analysis applying settings outlined in the latest study was used to calculate the appropriate sample size, with the results indicating that 60 participants per group (intervention and control group) would provide a sufficiently large Cohen's d effect size.

INSTRUMENTS AND DATA COLLECTION

Intervention: The blended learning module and online learning module for mentoring education for interprofessional dental health care professionals.

Instruments: Mentors' Competence in mentoring will be measured using the self-assessment of the Mentors' Competence Instrument (MCI), which includes seven mentoring competence sub-dimensions and 45 items.

Finnish language versions of the questionnaire will contain the following sections:

1. Sociodemographic data:

   * Sex
   * Age
   * Education background
   * Year of completion of education
   * Job title
   * Place of work
   * Work experience
   * Role of mentor
   * A time when last mentored a student
   * A most recent case of mentoring
   * Previous participation to mentoring education
   * Experience of previous mentoring education
2. Competence in mentoring using MCI, which contains 45 items divided into 7 sections

   * mentor characteristics
   * mentor motivation
   * mentoring practices in the workplace
   * reflection during mentoring
   * goal-oriented mentoring
   * student-centered evaluation
   * constructive feedback

DATA COLLECTION

Intervention group

1. Blended learning approach to mentoring education for dental health care professionals; Baseline questionnaire (T0): Paper-based questionnaires will be administered to participants in the intervention group on the day of study recruitment before mentoring education. A researcher will provide details to participants on the completion of the questionnaire.

   The online mentoring education (T0): Online questionnaire will be administered to participants in the intervention group by giving a weblink with the cover letter of the questionnaire outlines to the study purpose, protecting participant anonymity, and contact details of the researchers.
2. Post-course questionnaire (T1): A blended learning approach to mentoring education for dental health care professionals; Paper-based questionnaires will be administered to participants in the intervention group immediately following completion of the mentoring education.

   The interprofessional online mentoring education (T1): Online questionnaire will be administered to participants in the intervention group immediately following completion of the mentoring education.
3. Follow-up of the 3-month questionnaire (T2): A blended learning approach to mentoring education for dental health care professionals; Paper-based questionnaires will be sent to participants via post to participants' home addresses. The online mentoring education; An online questionnaire will be sent to weblink to participants via participants' email.

Control group

1. Baseline questionnaire (T0): Paper-based questionnaires will be sent in sealed envelop to participants of the control group during the timeline of the intervention group's mentoring education.
2. Post questionnaire (T1): Paper-based questionnaires will be sent in sealed envelop to participants of the control group after five weeks of the baseline measurement.
3. Follow-up of the 3-month questionnaire (T2): Paper-based questionnaire will be sent in sealed envelop to participants of the control group after three months of the baseline measurement.

ETHICAL CONSIDERATIONS

All phases of the study will follow guidelines for ethical research. The study will not require a statement from the ethics committee, as the research will not violate the participants' physical integrity and/or cause physical or mental harm. Permission for data collection was obtained from the organizations where education will be conducted. Participants will be informed of the study's purpose, the voluntary of their participation and of their right to withdraw from the study, protection of participants' anonymity, and contact details of the researchers. Answering the questionnaire was taken as an informed agreement to participate in the study. All of the collected data will be coded according to the key code in questionnaires T1, T2 and T2. The results of the study will be reported according to the CONSORT 2010 Statement and the TIDieR checklist. Process evaluations of the designed interventions will be reported in accordance with the Medical Research Council (MRC) guidelines. Respondent confidentiality will be assured throughout the study.

Data analysis

Data will be analyzed with SPSS (V. 22.0, IBM Corporation, Armonk, NY). Data will be analyzed using descriptive statistics, the Mann-Whitney U test and pre-and post-test changes will be assessed using the Wilcoxon Signed-Rank test. Parametric data analysis methods will be used for sensitivity testing. In this study, will be used two-tailed testing and the significance level will be set at a p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Dentist or dental hygienist
* Working in dental health care
* Readiness to participate in the study.

Exclusion Criteria:

* Professional from a field other than dental health care
* Unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Competence in mentoring students in the clinical practice | The Outcome Measures will be assessed a change. The change is being assessed; Pre intervention, immediately after intervention and 3 months after intervention.
  Mentor competence will be measured using the Mentors' Competence Instrument (MCI), which includes seven sum-variables and 45 items. Respondents rate each item of the instrument using a four-point Likert scale.(1=totally disagree, 2=disagree to some extent, 3=agree to some extent, and 4=totally agree). Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Changes in mentoring students | The Outcome Measures will be assessed a change. The change is being assessed; Immediately after intervention and 3 months after intervention.
  Satisfaction with mentoring education. The willingness of mentoring student. Measured will be using the Mentors' Competence Instrument (MCI), which includes seven sum-variables and 45 items. Respondents rate each item of the instrument using a four-point Likert scale. (1=totally disagree, 2=disagree to some extent, 3=agree to some extent, and 4=totally agree). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Mikkonen, PhD, Study Chair — University of Oulu; Anna-Leena Keinänen, MHSc, Principal Investigator — University of Oulu. Oulu University of Applied Sciences
Locations (1):
- Healthcare organizations in Nordic Finland, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilbert JH, Yan J, Hoffman SJ. A WHO report: framework for action on interprofessional education and collaborative practice. J Allied Health. 2010 Fall;39 Suppl 1:196-7. PMID 21174039
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] Keinanen AL, Mikkonen K, Lahdesmaki R, Kaariainen M. The dental healthcare professionals' competence in mentoring students in the clinical practice. Eur J Dent Educ. 2021 May;25(2):385-396. doi: 10.1111/eje.12615. Epub 2020 Oct 30. PMID 33058327
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] Rasanen L, Moore E. Critical evaluation of the guidelines of the Finnish Advisory Board on Research Integrity and of their application. Res Integr Peer Rev. 2016 Oct 17;1:15. doi: 10.1186/s41073-016-0020-9. eCollection 2016. PMID 29451531
- [Background] Tuomikoski AM, Ruotsalainen H, Mikkonen K, Miettunen J, Juvonen S, Sivonen P, Kaariainen M. How mentoring education affects nurse mentors' competence in mentoring students during clinical practice - A quasi-experimental study'. Scand J Caring Sci. 2020 Mar;34(1):230-238. doi: 10.1111/scs.12728. Epub 2019 Jun 28. PMID 31250935
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714